CLINICAL TRIAL: NCT01914653
Title: SERI® Surgical Scaffold Postmarket Study of Soft Tissue Support and Repair in Breast Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sofregen Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SURE-006
Record Dates: First submitted 2013-07-31; First posted 2013-08-02 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Breast Reconstruction

ARMS (3):
- Pre-radiated (Experimental)
  Interventions: Device: Silk surgical mesh
- Not radiated (Experimental)
  Interventions: Device: Silk surgical mesh
- Post-radiated (Experimental)
  Interventions: Device: Silk surgical mesh

INTERVENTIONS:
Device: Silk surgical mesh — A CE Marked, 510(k) cleared, knitted, multi-filament, bioengineered, silk mesh indicated for use as a transitory scaffold for soft tissue support and repair

SUMMARY:
Prospective, single center, postmarket clinical study to obtain clinical experience with the use of SERI® Surgical Scaffold for soft tissue support and repair in breast reconstruction.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for enrollment, the subject must:

1. Be female, ≥ 18 years of age
2. If the subject is a female of childbearing potential, have a pregnancy test evaluated as negative prior to surgery, per the site's standard of care
3. Have a nicotine test evaluated as negative prior to surgery and agree not to smoke for the duration of the study
4. Be willing to undergo mastectomy with healthy, well-vascularized skin flaps anticipated by the surgeon
5. Be eligible to enroll in one of the following three cohorts:

1. Subject had radiation therapy (XRT) prior to direct-to-implant (DTI) reconstruction, but will not have XRT following reconstruction;

2. Subject did not have XRT prior to DTI reconstruction and will not have XRT following reconstruction;

3. Subject did not have XRT prior to DTI reconstruction, but will have XRT following reconstruction.

Exclusion Criteria:

To be eligible for enrollment, the subject must not:

1. Have collagen-vascular, connective tissue, or bleeding disorders
2. Have any disease, including uncontrolled diabetes, which is clinically known to impact wound healing ability
3. Have an autoimmune disease, an immune deficiency, or is on immune-suppression drugs for reasons other than current treatment for breast cancer
4. Have a BMI that is ≥ 32
5. Have a nicotine test evaluated as positive prior to surgery or unwilling to quit smoking for the duration of the study
6. Currently have an alcohol/substance abuse problem or have had a relapse within 1 year prior to screening visit
7. Be pregnant, lactating, or expecting to be within the next 24 months
8. Have concomitant unrelated condition of breast/chest wall/skin (e.g. significant chest wall abnormalities including pectus excavatum or pectus carinatum)
9. Require the use of any additional implant for soft tissue support of the contralateral non-study breast, except in bilateral breast reconstructions, where the use of SERI® Surgical Scaffold is allowed
10. Have had a prior soft tissue support implant
11. If enrolled into the Pre-Radiated cohort, have had recent radiation (< 1 year) to the breast/chest wall
12. If enrolled into the Post-Radiated cohort, radiation to the breast/chest wall is planned more than 1 year from the time of SERI® Surgical Scaffold placement
13. Have clinical evidence of severe radiation tissue damage (e.g. pigmentation, indentation, atrophy, no elasticity to skin of radiated breast) from previous XRT to the breast/chest wall
14. Have large or multiple scars on the breast(s) that may interfere with blood supply to the mastectomy flaps

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Incidence of Implant Loss | 24 months postoperatively
  Implant Loss will be defined as situations in which the breast implant is removed and not immediately replaced.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan Medical
Locations (1):
- Assuta Medical Center, Tel Aviv, Israel